CLINICAL TRIAL: NCT05099510
Title: A Phase I Open Label, Placebo-controlled Dose Escalation Study to Evaluate Safety and Pharmacokinetics of NatrunixTM Via Subcutaneous Injection in Healthy Subjects
Brief Title: Natrunix Safety PK Study in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: XBiotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-PT053
Record Dates: First submitted 2021-09-16; First posted 2021-10-29 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Each subject will receive a single subcutaneous injection of Natrunix at one of the three doses (200 mg, 400 mg or 800 mg) or placebo. For each dose cohort, six subjects will be administered Natrunix and two subjects will be administered placebo. The study will not proceed to the next dose level unless the tested dose level has been deemed to have acceptable tolerability and safety. Subjects will undergo blood sampling for toxicity and pK analysis. Subjects will also be evaluated for the development of anti-drug antibodies (ADA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NatrunixTM (Active Comparator): Each participant will receive one single subcutaneous injection of 200 mg (Cohort 1), 400 mg (Cohort 2), or 800 mg (Cohort 3) of NatrunixTM.
  Interventions: Biological: NatrunixTM
- Placebo (Placebo Comparator): Each participant will receive one single subcutaneous injection of placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NatrunixTM — The active ingredient in the drug product NatrunixTM is XB2001, a recombinant human IgG4 monoclonal antibody specific for human interleukin-1-alpha (IL-1-alpha). The entire XB2001 heavy and light chain sequences are identical to those found in naturally-occurring human IgG4-kappa, with the light and heavy chain variable regions being identical to those originally expressed by a peripheral blood B lymphocyte that was obtained from a healthy individual.
  Arms: NatrunixTM
Biological: Placebo — Placebo control for NatrunixTM subcutaneous injection.
  Arms: Placebo

SUMMARY:
This trial will be a Phase I Open Label, Placebo-controlled Dose Escalation Study to Evaluate Safety and Pharmacokinetics of Natrunix via Subcutaneous Injection in Healthy Subjects. The target enrollment is 8 healthy subjects per cohort (including six for Natrunix and two for placebo). Three cohorts for a total of 24 healthy volunteers.

DETAILED DESCRIPTION:
Study Title: A Phase I Open Label, Placebo-controlled Dose Escalation Study to Evaluate Safety and Pharmacokinetics of Natrunix via Subcutaneous Injection in Healthy Subjects.

Sponsor: XBiotech USA, Inc.

Study Chair: Neha Reshamwala, MD

Number of Planned Subjects: Eight healthy subjects per cohort (including six for Natrunix and two for placebo). Three cohorts for a total of 24 healthy volunteers.

Approximate Duration: Approximately 38 days for each subject which includes a screening period of up to 10 days followed by one subcutaneous dose of Natrunix, and then evaluation over 28 days. Blood will be sampled at various time points for blood chemistry, hematological analysis and Natrunix serum/plasma concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18
2. Adequate bone marrow function defined as:

   * absolute neutrophil count (neutrophil and bands) of ≥ 1,500/mm3 (≥ 1.5 x 109/L)
   * platelet count > 150,000/mm3
   * hemoglobin of ≥ 10 g/dL
3. Adequate renal function, defined by serum creatinine ≤ 1.5 x lab ULN.
4. Adequate hepatic function defined as:
5. serum albumin ≥ 3.0 g/dL
6. total bilirubin ≤ 1.5 times lab ULN.
7. alanine aminotransferase (ALT) ≤ 2.0 times lab ULN.
8. aspartate aminotransferase (AST) ≤ 2.0 times lab ULN
9. For WOCBP, a negative pregnancy test at screening. For subjects with reproductive potential, willingness to use one method of contraception of high efficacy during the entire study period. These methods can include but not limited to hormonal contraceptives, intrauterine devices, condoms, diaphragms etc. Women of non-childbearing potential include those considered to have a medical history that indicates that pregnancy is not a reasonable risk, including post-menopausal women and those with a history of hysterectomy or surgically sterilized.
10. If the participant is a male participating in this clinical research study, the subject should not get a sexual partner pregnant during participation in this research study as the effect of the study drug on sperm is not known. The male contraception methods can include but not limited to mechanical methods (abstinence, withdrawal, non-vaginal intercourse) or contemporary methods comprising condoms and vasectomy.
11. Signed and dated Institutional Review Board (IRB) approved informed consent before any protocol-specific screening procedures are performed.

Exclusion Criteria:

1. Treatment with any biologicals (including intravenous immunoglobulin) or investigational agents within the last 4 weeks (or 5 half-lives, whichever is longer).
2. Uncontrolled or significant cardiovascular disease, including:

   * A myocardial infarction within the past 6 months.
   * Uncontrolled angina within the past 3 months.
   * Congestive heart failure within the past 3 months, defined as New York Heart Association (NYHA) Class II or higher.
   * Uncontrolled hypertension (blood pressure >160 mm Hg systolic or >100 mm Hg diastolic).
3. Dementia or altered mental status that would prohibit the understanding or rendering of informed consent.
4. Treatment with immunosuppressant agents, including corticosteroids or cyclosporine within the last 4 weeks.
5. Serious uncontrolled medical disorders, such as uncontrolled diabetes, active peptic ulcer disease, cerebrovascular accident within three months, ongoing congestive heart failure, and any other condition, which in the opinion of the investigator, would put the subject at risk by participating in the trial.
6. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
7. Abnormal ECG with any clinically significant findings or with QTc > 470 ms.
8. Infection requiring treatment with antibiotics within 3 weeks prior to screening.
9. Infectious disease:

   • Positive HIV, RPR, Hepatitis B or C, TB (QuantiFERON-TB Gold (QFT)/ IGRA)
10. History of immunodeficiency.
11. Female subjects who are pregnant, planning to become pregnant during the course of the study, or breast-feeding.
12. Major surgery within 28 days prior to Day 0.
13. History of progressive multifocal leukoencephalopathy (PML) or other demyelinating disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with treatment related adverse events assessed according to CTCAE v5.0 | 28 days
  Participants will be monitored for acute reactions, blood chemistry and hematology immediately after dosing and at multiple time points up to 28 days. All adverse events will be documented at multiple time points and assessed in terms those possibly, probably and definitely related to test article according to CTCAE v4.0 criteria. Anti-drug antibodies (ADA) will also be evaluated.

SECONDARY OUTCOMES:
Maximum plasma concentration of test article 2) Terminal plasma concentration 3) Plasma half-life 4) Total exposure | 28 days
  The maximum plasma concentration will be assessed using a proprietary immunoassay to detect circulating NatrunixTM
Terminal plasma concentration | 28 days
  Terminal plasma concentration will be assessed at 28 days.
Half-life | 28 days
  Peak and terminal plasma levels will be used in a two compartmental model to assess plasma half-life.
Total exposure | 28 days
  Area under the curve will be determined based on measured plasma levels over 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Reshamwala, MD, Principal Investigator — BioBehavioral Research of Austin
Locations (1):
- BioBehavioral Research of Austin, A Telemed2U Company, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No It is not yet known if there will be a plan to make IPD available